CLINICAL TRIAL: NCT02444364
Title: Pilot Project Evaluation of the DPP-4 Inhibition With Sitagliptin on Calcium and Bone Metabolism in Patients With Type 2 Diabetes Mellitus
Brief Title: Effects of DPP-4 Inhibition on Calcium and Bone Metabolism in Type 2 Diabetes Mellitus
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Funding withdrawn; no participants enrolled.
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MERCK-200379
Record Dates: First submitted 2015-05-11; First posted 2015-05-14 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; bone loss; Bone Density
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Bone Diseases, Metabolic | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sitagliptin (Experimental): Subjects will receive 90 tablets of 100mg sitagliptin
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Sitagliptin — Subjects will receive 90 tablets of 100mg sitagliptin
  Other Names: Januvia

SUMMARY:
Participants will be persons with Type 2 Diabetes who are likely to have increased risk of bone fractures. The investigators believe this medication will enhance bone turnover.

The investigators will use DXA measurements to evaluate bone density before and after subjects take the medication.

DETAILED DESCRIPTION:
Type 2 Diabetes Mellitus (T2DM) is associated with an increased risk of bone fractures even when there is not decreased bone density via DXA measurements. This appears primarily related to impaired bone quality and abnormal bone architecture. Although the exact pathophysiologic mechanisms remain unclear, low bone turnover is considered one of the key defects. Emerging evidence suggests that dipeptidyl peptidase (DPP) inhibition is associated with improved bone quality and reduction in fracture risk.

While animal studies have shown an improvement in bone mineral density and trabecular architecture with sitagliptin treatment, no such studies in humans have yet been undertaken. We are proposing to extend these animal studies with a pilot clinical trial that seeks to use serum markers of bone turn-over and calcaneal quantitative ultrasound to evaluate the effect of DPP-4 inhibition on bone metabolism. Our hypothesis is that DPP-4 inhibition with sitagliptin will enhance bone turn over and quality in persons with T2DM.

This project project seeks to examine the impact of six months of therapy on sitagliptin, a DPP-4 inhibitor, on bone metabolism and bone quality in subjects with T2DM. The proposed study is intended to be a pilot investigation for providing preliminary data for submission of a more definitive national grant proposal with a larger patient population, blinded randomized control design and high resolution CT imaging of the lumbar spine.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes mellitus.
2. Hemoglobin A1c >6.5% and <10%.
3. Estimated GFR greater than 60 mL per minute per meter squared.
4. Between 18 and 70 years of age.
5. On oral antihyperglycemic agents with stable dose at least for last 2 months.
6. Females: minimum of two years postmenopausal, surgically sterile, or using an acceptable contraceptive regimen (OCP, IUD, double barrier, Depo-Provera or subcutaneous progestin implant) and negative urine pregnancy test at trial start.

Exclusion Criteria:

1. Pregnancy, breast feeding or planning pregnancy during the study period
2. Any medical condition expected to be terminal within one year
3. Active mental illness or other condition which in the opinion of the investigator would prevent informed consent or adherence with study protocol
4. Use of any PPAR agonist within three months prior to enrollment
5. Daily insulin use
6. Vitamin D level < 20
7. Allergy or intolerance of sitagliptin or other DPP-4 inhibitor
8. Use of DPP-4 inhibitor or GLP-1 analog within three months prior to enrollment
9. Significant alcohol use defined as >3 standard servings of alcohol per day for men and >2 for women
10. History of bariatric surgery in the last 3 years or planned bariatric surgery during the study period
11. Receipt of another study drug within 30 days of screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in Bone Turnover | Six Months

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed T Sarmini, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia: Diabetes Center, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No